CLINICAL TRIAL: NCT04728100
Title: Smartphone and Smartwatch Based ECG for Patients With Congenital Long QT Syndrome
Brief Title: LQT and Smartphone/Smartwatch
Acronym: SMART-QT
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL20_1052
Record Dates: First submitted 2021-01-21; First posted 2021-01-28 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Long QT Syndrome
MeSH Terms: conditions — Long QT Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: LQT — Patients with LQT syndrome diagnosis.

SUMMARY:
Congenital long QT syndrome (LQTS) is a rare genetic disorder characterized by prolongation of the corrected QT interval (QTc) on the electrocardiogram. LQTS is associated with a risk of syncope or sudden death from ventricular arrhythmia.

The increase in the duration of the corrected QT interval and / or changes in the morphology of the T wave on the electrocardiogram are markers of an increased risk of sudden death and syncope.

Recently, a personal portable 6-lead device (DI, DII, DIII, aVF, aVL and aVR) connected to the patient's smartphone has entered the market (KARDIA MOBILE 6L, AliveCor, Mountain View, CALIFORNIA, USA). The APPLE WATCH Series 6 (Apple, Cupertino, CA, USA) can also record an ECG. If the device is designed to record a single lead (DI), several works have shown that it is possible to record 9 leads (DI, DII, DIII, V1, V2, V3, V4, V5 and V6) by moving simply the device (Spaccarotella CAS et al. JAMA Cardiology 2020).

These devices were originally designed to screen for atrial fibrillation, but they produce accurate 6- and 9-lead ECGs and could potentially allow ambulatory ECG monitoring of patients with LQTS.

ELIGIBILITY:
Inclusion Criteria:

Patient with diagnosis of LQTS based on the following criteria:

* Corrected QT (Qtc) interval according to Bazett method ≥ 480 ms, at several times in the absence of a secondary cause
* and / or class 4 or 5 mutation in a gene involved in long QT syndrome
* and / or syncope (s) and QTc> 460ms in the absence of other cause

  * All ages
  * No opposition from the patient

Exclusion Criteria:

None

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: LQT patients
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

PRIMARY OUTCOMES:
the duration of the QTc (ms) | at the inclusion visit
  The primary outcome is the measurement of 3 data:
  - the duration of the QTc (ms). These data will be measured during the same inclusion visit with 1/ the standard 12-lead ECG machine, 2/ the KARDIA MOBILE 6L and 3/the APPLE WATCH Series 6. The data of the Kardia Mobile 6L and the Apple Watch series 6 will be compared to the data of the gold standard a 12-lead ECG.
the morphology of the T waves (bpm). | at the inclusion visit
  - the morphology of the T waves (bpm). These data will be measured during the same inclusion visit with 1/ the standard 12-lead ECG machine, 2/ the KARDIA MOBILE 6L and 3/the APPLE WATCH Series 6. The data of the Kardia Mobile 6L and the Apple Watch series 6 will be compared to the data of the gold standard a 12-lead ECG.
the heart rate (bpm). | at the inclusion visit
  - the heart rate (bpm). These data will be measured during the same inclusion visit with 1/ the standard 12-lead ECG machine, 2/ the KARDIA MOBILE 6L and 3/the APPLE WATCH Series 6. The data of the Kardia Mobile 6L and the Apple Watch series 6 will be compared to the data of the gold standard a 12-lead ECG.

CONTACTS AND LOCATIONS:
Locations (1):
- Chevalier, Bron, France

REFERENCES:
- [Derived] Deliniere A, Bessiere F, Placide L, Pasquie JL, Haddad C, Tirel S, Mokhtar H, Morel E, Gardey K, Dulac A, Ditac G, Sacher F, Denjoy I, Chevalier P. Wearable electrocardiogram devices in patients with congenital long QT syndrome: The SMART-QT study. Arch Cardiovasc Dis. 2024 May;117(5):313-320. doi: 10.1016/j.acvd.2024.02.010. Epub 2024 Apr 24. PMID 38704288